CLINICAL TRIAL: NCT01939548
Title: A 12-week , Randomized, Phase 2, Double-blind, Parallel-group Study Of Two Dose Levels Of Pf-02545920 Compared To Placebo In The Adjunctive Treatment Of Outpatients With Sub-optimally Controlled Symptoms Of Schizophrenia
Brief Title: An Outpatient Study Of The Efficacy, Safety, And Tolerability Of PF-02545920 In The Adjunctive Treatment Of Sub-Optimally Controlled Symptoms of Schizophrenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A pre-planned interim analysis indicated the trial was unlikely to meet the pre-specified efficacy criteria. The decision was not based on any safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A8241019
Record Dates: First submitted 2013-08-09; First posted 2013-09-11 (Estimated); Results first posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Schizophrenia
Keywords: PF-02545920; schizophrenia; outpatient; safety; efficacy; suboptimal response
MeSH Terms: conditions — Schizophrenia | interventions — 2-((4-(1-methyl-4-pyridin-4-yl-1H-pyrazol-3-yl)phenoxy)methyl)quinoline; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PF-02545920 (5mg) (Experimental)
  Interventions: Drug: PF-02545920
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-02545920 (15mg) (Experimental)
  Interventions: Drug: PF-02545920

INTERVENTIONS:
Drug: PF-02545920 — PF-02545920 2 mg BID x 7 days, then 5 mg BID until the Week 12 visit
  Other Names: 5 mg BID
  Arms: PF-02545920 (5mg)
Drug: Placebo — Placebo BID until the Week 12 visit
  Arms: Placebo
Drug: PF-02545920 — PF-02545920 5 mg BID x 7 days, then 10 mg BID x 7 days, then 15 mg BID until the Week 12 visit
  Other Names: 15 mg BID
  Arms: PF-02545920 (15mg)

SUMMARY:
This study aims to evaluate whether PF-02545920 is safe and effective in the treatment of sub-optimally controlled symptoms of schizophrenia during a 12-week outpatient treatment period. The study will use the Positive and Negative Syndrome Scale (PANSS) to measure change in symptoms for PF-02545920 from baseline compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatrically stable subjects with schizophrenia who have had a suboptimal response to current treatment
* Evidence of stable schizophrenia symptomatology greater than or equal to 3 months.
* Subjects must be on a stable medication treatment regimen greater than or equal to 2 months, including concomitant psychotropic medications.

Exclusion Criteria:

* History of seizures or of a condition with risk of seizures.
* Subjects with schizophrenia that have not responded at all to current treatment.
* Pregnant or nursing females, and females of child bearing potential.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- United States (44):
  - Birmingham Psychiatry Pharmaceutical Studies, Inc., Birmingham, Alabama
  - Woodland International Research Group, INC, Little Rock, Arkansas
  - Comprehensive Clinical Development, Inc., Cerritos, California
  - ProScience Research Group, Culver City, California
  - Synergy Clinical Research of Escondido, Escondido, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Pacific Research Partners, Oakland, California
  - Excell Research, Inc., Oceanside, California
  - Neuropsychiatric Research Center of Orange County, Orange, California
  - CiTrials, Riverside, California
  - CNRI-San Diego, LLC, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Collaborative Neuroscience Network, Inc., Torrance, California
  - Bliss Basement Pharmacy, Hartford, Connecticut
  - Institute of Living, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Comprehensive Clinical Development, Washington D.C., District of Columbia
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Florida Clinical research Center, LLC, Brandenton, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Medical Research Group of Central Florida, Sanford, Florida
  - Comprehensive Clinical Development, Inc., Atlanta, Georgia
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Chinmay K. Patel, DO, Hoffman Estates, Illinois
  - Behavioral Health Care Associates, Schaumburg, Illinois
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Louisiana Clinical Research, Shreveport, Louisiana
  - CBH Health, LLC, Rockville, Maryland
  - Psychiatric Care & Research Center, O'Fallon, Missouri
  - St. Louis Clinical Trials/The Summit@Creve Coeur, St Louis, Missouri
  - Altea Research, Las Vegas, Nevada
  - Comprehensive Clinical Development, Jamaica, New York
  - Manhattan Psychiatric Center's 125th St. Clinic, New York, New York
  - Manhattan Psychiatric Center, Ward's Island, New York
  - Midwest Clinical Research Center, LLC, Dayton, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - Community Clinical Research, Inc, Austin, Texas
  - Futuresearch Trials of Dallas, Dallas, Texas
  - Pillar Clinical Research LLC, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Psychiatric and Behaviorial Solutions, Salt Lake City, Utah
  - Lifetree Clinical Research, Salt Lake City, Utah

REFERENCES:
- [Derived] Targum SD, Cara Pendergrass J, Toner C, Zumpano L, Rauh P, DeMartinis N. Impact of BPRS interview length on ratings reliability in a schizophrenia trial. Eur Neuropsychopharmacol. 2015 Mar;25(3):312-8. doi: 10.1016/j.euroneuro.2014.11.023. Epub 2014 Dec 13. PMID 25554563
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8241019&StudyName=An%20Outpatient%20Study%20Of%20The%20Efficacy%2C%20Safety%2C%20And%20Tolerability%20Of%20PF-02545920%20In%20The%20Adjunctive%20Treatment%20Of%20Sub-Optimally%20Controlled%20S

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-02545920 5 mg BID: Participants received 1 placebo tablet and 2 PF-02545920 1 mg tablets twice daily (BID) from Days 1-7, followed by 2 placebo tablets and 1 PF-02545920 5 mg tablet BID from Days 8-84 (treatment phase). Study drug was self-administered orally BID by the participants based on instructions given at the sites. Participants took a total of 6 tablets per day (3 each in the morning and evening).
- PF-02545920 15 mg BID: Participants received 2 placebo tablets and 1 PF-02545920 5 mg tablet twice daily (BID) from Days 1-7, followed by 1 placebo tablet and 2 PF-02545920 5 mg tablets BID from Days 8-14 (treatment phase), and finally 3 PF-02545920 5 mg tablets from Days 15-84 (treatment phase). Study drug was self-administered orally BID by the participants based on instructions given at the sites. Participants took a total of 6 tablets per day (3 each in the morning and evening).
- Placebo: Participants received 3 placebo tablets from Days 1-84 (treatment phase). Study drug was self-administered orally BID by the participants based on instructions given at the sites. Participants took a total of 6 tablets per day (3 each in the morning and evening).
Period: Overall Study
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Started | 78 | 82 | 80
Completed | 41 | 33 | 50
Not Completed | 37 | 49 | 30
Not completed — Non compliance | 0 | 2 | 0
Not completed — Study Terminated by Sponsor | 17 | 19 | 12
Not completed — Insufficient Clinical Response | 1 | 0 | 0
Not completed — Did Not Meet Entrance Criteria | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 1
Not completed — Protocol Violation | 7 | 6 | 5
Not completed — Lost to Follow-up | 5 | 5 | 3
Not completed — Adverse Event | 2 | 9 | 7
Not completed — Death | 0 | 0 | 1
Not completed — Participant dropped | 0 | 0 | 1
Not completed — Participant unwilling to continue | 0 | 1 | 0
Not completed — Participant withdrew consent | 0 | 2 | 0
Not completed — Did not complete follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received study treatment were included in the baseline characteristics summary.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo | Total
Number analyzed (Participants) | 78 | 82 | 80 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (10.4) | 46.3 (9.4) | 45.6 (9.9) | 46.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 27 | 76
  Male | 55 | 56 | 53 | 164

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Syndrome Scale (PANSS) Total Score at Baseline
Description: The Positive and Negative Syndrome Scale (PANSS) assesses the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS Total Score and ranges from 30 to 210; higher score indicates greater severity.
Time Frame: Baseline
Population: All participants who received study treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 82 | 80
units on a scale | 81.7 (11.66) | 82.5 (11.71) | 80.8 (11.19)

2. Primary Outcome: Change From Baseline to Week 12 in PANSS Total Score
Description: The PANSS assesses the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS Total Score and ranges from 30 to 210; higher score indicates greater severity.
Time Frame: Baseline, Week 12
Population: All participants in the Full Analysis Set (FAS, defined as all participants who received at least 1 dose of randomized study medication, had a baseline and at least 1 post-baseline measurement) who had available data for this outcome measure at Week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 40 | 33 | 49
units on a scale | -13.1 (12.68) | -16.0 (13.76) | -16.7 (13.68)
Statistical Analysis 1: Comparison: PF-02545920 5 mg BID vs Placebo; Linear mixed-effect repeated measures model used. Fixed effects: treatment, time (visit), PANSS Total baseline value, investigator site; random effect: participant. Also included effects for treatment by time interaction and baseline value of PANSS Total by treatment interaction and background antipsychotics; Test type: Superiority or Other; p = 0.1991, Mixed Models Analysis — Primary analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; Least Squares Mean (LSM) Difference = 3.11, 80% CI 2-sided [0.01 to 6.21], Standard Error of Mean 2.409 — The estimation method used was restricted maximum likelihood
Statistical Analysis 2: Comparison: PF-02545920 15 mg BID vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3488, Mixed Models Analysis — Primary analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 2.30, 80% CI 2-sided [-0.85 to 5.45], Standard Error of Mean 2.445 — The estimation method used was restricted maximum likelihood

3. Secondary Outcome: Change From Baseline to Week 12 in Personal and Social Performance Scale (PSP) Total Score
Description: The Personal and Social Performance Scale (PSP) is a validated clinician-related scale that measured personal and social functioning in the domains of: socially useful activities (eg, work and study), personal and social relationships, self-care, disturbing and aggressive behaviors. Information from the participant and the informant were utilized in determining the rating. A PSP total score was determined from the 4 domains (score range 0-100). A score between 71 and 100 indicates a mild degree of difficulty; a score between 31 and 70 indicates a moderate degree of dysfunction, and a participant with a score of 30 or less has functioning so poor he or she requires intensive supervision.
Time Frame: Baseline, Week 12
Population: All participants who received study treatment were included in the baseline evaluation. The number of evaluable participants at Week 12 were those in the FAS with available data at Week 12 (n=number of evaluable participants at the specified time point)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 82 | 80
units on a scale
  Baseline (n=78, 82, 80) | 54.3 (9.14) | 53.9 (10.38) | 52.6 (10.18)
  Change at Week 12 (n=40, 34, 50) | 6.3 (7.25) | 6.0 (10.12) | 8.7 (10.19)
Statistical Analysis 1: Comparison: PF-02545920 5 mg BID vs Placebo; Analysis of change at Week 12. Linear mixed-effect repeated measures model used. Fixed effects: treatment, time (visit), baseline value, investigator site; random effect: participant. Also included effects for treatment by time interaction and baseline value by treatment interaction and background antipsychotics; Test type: Superiority or Other; p = 0.8786, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = -0.23, 80% CI 2-sided [-2.13 to 1.67], Standard Error of Mean 1.476 — The estimation method used was restricted maximum likelihood
Statistical Analysis 2: Comparison: PF-02545920 15 mg BID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.4483, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = -1.14, 80% CI 2-sided [-3.08 to 0.79], Standard Error of Mean 1.502 — The estimation method used was restricted maximum likelihood

4. Secondary Outcome: Change From Baseline to Week 12 in PANSS Positive, Negative, and General Subscales
Description: The PANSS includes 3 scales and 30 items: 7 items that make up the Positive Scale (eg, delusions, conceptual disorganization, hallucinatory behavior); 7 items that make up the Negative Scale (eg, blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal); and 16 items that make up the General Psychopathology Scale (eg, somatic concern, anxiety, guilt feelings, mannerisms and posturing, motor retardation, uncooperativeness, disorientation, poor impulse control, preoccupation). Individual items are scored with values ranging from 1 to 7. Total Negative and Positive Subscale scores each range from 7 to 49; higher score indicates greater severity. Total General Psychopathology Subscale score range from 16 to 112; higher score indicates greater severity.
Time Frame: Baseline, Week 12
Population: All participants who received study treatment were included in the baseline evaluation. At Week 12, the number of evaluable participants in the FAS were 40, 33, and 49.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 82 | 80
units on a scale
  Positive subscale score, baseline | 21.4 (4.05) | 21.3 (4.83) | 21.8 (4.07)
  Positive subscale score, change at Week 12 | -4.2 (3.91) | -3.6 (4.34) | -5.3 (4.25)
  Negative subscale score, baseline | 20.5 (4.01) | 20.6 (4.27) | 20.6 (4.30)
  Negative subscale score, change at Week 12 | -3.0 (4.22) | -3.6 (4.90) | -3.7 (4.13)
  General subscale score, baseline | 39.8 (6.96) | 40.7 (6.79) | 38.4 (6.02)
  General subscale score, change at Week 12 | -6.0 (7.23) | -8.8 (7.94) | -7.7 (7.69)
Statistical Analysis 1: Comparison: PF-02545920 5 mg BID vs Placebo; Positive Subscale Score comparison of change at Week 12. Linear mixed-effect repeated measures model used. Fixed effects: treatment, time (visit), baseline value, investigator site; random effect: participant. Also included effects for treatment by time interaction and baseline value by treatment interaction and background antipsychotics; Test type: Superiority or Other; p = 0.3201, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 0.81, 80% CI 2-sided [-0.23 to 1.85], Standard Error of Mean 0.809 — The estimation method used was restricted maximum likelihood
Statistical Analysis 2: Comparison: PF-02545920 15 mg BID vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.2961, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 0.85, 80% CI 2-sided [-0.19 to 1.90], Standard Error of Mean 0.813 — The estimation method used was restricted maximum likelihood
Statistical Analysis 3: Comparison: PF-02545920 5 mg BID vs Placebo; Negative Subscale Score comparison of change at Week 12. Linear mixed-effect repeated measures model used. Fixed effects: treatment, time (visit), baseline value, investigator site; random effect: participant. Also included effects for treatment by time interaction and baseline value by treatment interaction and background antipsychotics; Test type: Superiority or Other; p = 0.6015, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 0.39, 80% CI 2-sided [-0.57 to 1.35], Standard Error of Mean 0.743 — The estimation method used was restricted maximum likelihood
Statistical Analysis 4: Comparison: PF-02545920 15 mg BID vs Placebo; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.7787, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 0.21, 80% CI 2-sided [-0.77 to 1.19], Standard Error of Mean 0.761 — The estimation method used was restricted maximum likelihood
Statistical Analysis 5: Comparison: PF-02545920 5 mg BID vs Placebo; General Subscale Score comparison of change at Week 12. Linear mixed-effect repeated measures model used. Fixed effects: treatment, time (visit), baseline value, investigator site; random effect: participant. Also included effects for treatment by time interaction and baseline value by treatment interaction and background antipsychotics; Test type: Superiority or Other; p = 0.2068, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 1.63, 80% CI 2-sided [-0.02 to 3.29], Standard Error of Mean 1.285 — The estimation method used was restricted maximum likelihood
Statistical Analysis 6: Comparison: PF-02545920 15 mg BID vs Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.4611, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 0.98, 80% CI 2-sided [-0.73 to 2.69], Standard Error of Mean 1.326 — The estimation method used was restricted maximum likelihood

5. Secondary Outcome: Change From Baseline to Week 12 in PANSS-Derived Marder Factor Scores
Description: The subscales based on Marder factors are: negative symptoms, positive symptoms, disorganized thoughts factor, uncontrolled hostility/excitement factor, and anxiety/depression factor. The symptoms are rated on a 7-point scale, with a range of 7 to 49 for negative symptoms, 8 to 56 for positive symptoms, 7 to 49 for disorganized thoughts and 4 to 28 for uncontrolled hostility/excitement and anxiety/depression. Higher scores indicate higher severity of symptoms.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 82 | 80
units on a scale
  Anxiety/depression, baseline | 10.7 (3.16) | 10.9 (3.03) | 10.0 (2.95)
  Anxiety/depression, change at Week 12 (W12) | -1.9 (4.09) | -2.4 (3.71) | -2.9 (3.15)
  Disorganized thought, baseline | 17.4 (3.40) | 17.5 (4.11) | 17.5 (3.80)
  Disorganized thought, change at W12 | -2.4 (2.92) | -3.9 (3.25) | -2.2 (3.24)
  Negative symptom, baseline | 20.7 (4.44) | 20.8 (4.71) | 20.4 (4.62)
  Negative symptom, change at W12 | -3.4 (4.50) | -4.2 (5.19) | -4.4 (4.52)
  Positive symptom, baseline | 25.3 (4.72) | 24.9 (5.23) | 25.3 (4.90)
  Positive symptom, change at W12 | -4.6 (4.71) | -3.6 (5.49) | -5.5 (4.61)
  Uncontrolled hostility/excitement, baseline | 7.7 (2.58) | 8.5 (2.96) | 7.5 (2.65)
  Uncontrolled hostility/excitement, change at W12 | -0.8 (2.22) | -1.9 (2.25) | -1.6 (2.76)
Statistical Analysis 1: Comparison: PF-02545920 5 mg BID vs Placebo; Anxiety/depression symptom score comparison of change at Week 12. Linear mixed-effect repeated measures model used. Fixed effects: treatment, time (visit), baseline value, investigator site; random effect: participant. Also included effects for treatment by time interaction and baseline value by treatment interaction and background antipsychotics; Test type: Superiority or Other; p = 0.1083, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 0.96, 80% CI 2-sided [0.19 to 1.72], Standard Error of Mean 0.591 — The estimation method used was restricted maximum likelihood
Statistical Analysis 2: Comparison: PF-02545920 15 mg BID vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0869, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 1.05, 80% CI 2-sided [0.27 to 1.84], Standard Error of Mean 0.611 — The estimation method used was restricted maximum likelihood
Statistical Analysis 3: Comparison: PF-02545920 5 mg BID vs Placebo; Disorganized thought symptom score comparison of change at Week 12. Linear mixed-effect repeated measures model used. Fixed effects: treatment, time (visit), baseline value, investigator site; random effect: participant. Also included effects for treatment by time interaction and baseline value by treatment interaction and background antipsychotics; Test type: Superiority or Other; p = 0.8601, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = -0.10, 80% CI 2-sided [-0.84 to 0.64], Standard Error of Mean 0.575 — The estimation method used was restricted maximum likelihood
Statistical Analysis 4: Comparison: PF-02545920 15 mg BID vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p = 0.3454, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = -0.56, 80% CI 2-sided [-1.33 to 0.20], Standard Error of Mean 0.593 — The estimation method used was restricted maximum likelihood
Statistical Analysis 5: Comparison: PF-02545920 5 mg BID vs Placebo; Negative symptom score comparison of change at Week 12. Linear mixed-effect repeated measures model used. Fixed effects: treatment, time (visit), baseline value, investigator site; random effect: participant. Also included effects for treatment by time interaction and baseline value by treatment interaction and background antipsychotics; Test type: Superiority or Other; p = 0.3273, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 0.78, 80% CI 2-sided [-0.24 to 1.79], Standard Error of Mean 0.789 — The estimation method used was restricted maximum likelihood
Statistical Analysis 6: Comparison: PF-02545920 15 mg BID vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.3963, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 0.69, 80% CI 2-sided [-0.35 to 1.72], Standard Error of Mean 0.806 — The estimation method used was restricted maximum likelihood
Statistical Analysis 7: Comparison: PF-02545920 5 mg BID vs Placebo; Positive symptom score comparison of change at Week 12. Linear mixed-effect repeated measures model used. Fixed effects: treatment, time (visit), baseline value, investigator site; random effect: participant. Also included effects for treatment by time interaction and baseline value by treatment interaction and background antipsychotics; Test type: Superiority or Other; p = 0.4713, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 0.64, 80% CI 2-sided [-0.50 to 1.78], Standard Error of Mean 0.888 — The estimation method used was restricted maximum likelihood
Statistical Analysis 8: Comparison: PF-02545920 15 mg BID vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.1787, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 1.21, 80% CI 2-sided [0.06 to 2.36], Standard Error of Mean 0.895 — The estimation method used was restricted maximum likelihood
Statistical Analysis 9: Comparison: PF-02545920 5 mg BID vs Placebo; Uncontrolled hostility/excitement symptom score comparison of change at Week 12. Linear mixed-effect repeated measures model used. Fixed effects: treatment, time (visit), baseline value, investigator site; random effect: participant. Also included effects for treatment by time interaction and baseline value by treatment interaction and background antipsychotics; Test type: Superiority or Other; p = 0.4123, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 0.35, 80% CI 2-sided [-0.20 to 0.90], Standard Error of Mean 0.426 — The estimation method used was restricted maximum likelihood
Statistical Analysis 10: Comparison: PF-02545920 15 mg BID vs Placebo; [analysis description as in outcome 5, analysis 9]; Test type: Superiority or Other; p = 0.3202, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = -0.44, 80% CI 2-sided [-1.01 to 0.13], Standard Error of Mean 0.441 — The estimation method used was restricted maximum likelihood

6. Secondary Outcome: Change From Baseline to Week 12 in Clinical Global Impression of Severity (CGI-S)
Description: CGI-S: 7-point clinician-rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected. Change: score at observation minus score at baseline.
Time Frame: Baseline, Week 12
Population: All participants who received study treatment were included in the baseline evaluation. n=number of evaluable participants in the FAS at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 82 | 80
units on a scale
  Baseline (n=78, 82, 80) | 4.3 (0.50) | 4.3 (0.45) | 4.4 (0.54)
  Change at Week 12 (n=40, 34, 50) | -0.8 (0.78) | -0.7 (0.59) | -0.8 (0.74)
Statistical Analysis 1: Comparison: PF-02545920 5 mg BID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.7399, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 0.04, 80% CI 2-sided [-0.11 to 0.19], Standard Error of Mean 0.119 — The estimation method used was restricted maximum likelihood
Statistical Analysis 2: Comparison: PF-02545920 15 mg BID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2747, Mixed Models Analysis — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 0.13, 80% CI 2-sided [-0.02 to 0.29], Standard Error of Mean 0.122 — The estimation method used was restricted maximum likelihood

7. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Total Score at Week 12
Description: CGI-I: 7-point clinician-rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: Week 12
Population: Participants in the FAS who were evaluable for this outcome measure at Week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 40 | 34 | 50
units on a scale | 2.9 (1.00) | 2.7 (0.96) | 2.9 (0.88)
Statistical Analysis 1: Comparison: PF-02545920 5 mg BID vs Placebo; Analysis of change at Week 12. Mixed effect repeated measures model used. Fixed effects: treatment, time (visit), baseline value, investigator site, visit and visit-by-treatment interaction; random effect: participant; Test type: Superiority or Other; p = 0.7219, ANOVA — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = 0.07, 80% CI 2-sided [-0.17 to 0.31], Standard Error of Mean 0.188
Statistical Analysis 2: Comparison: PF-02545920 15 mg BID vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.9315, ANOVA — Analysis was two-sided and performed at the 0.2 significance level. No multiple comparisons adjustment was made; LSM Difference = -0.02, 80% CI 2-sided [-0.26 to 0.23], Standard Error of Mean 0.192

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Discontinuations Due to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. AEs comprised both SAEs and non-SAEs. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent adverse events (TEAEs) were defined as newly occurring AEs or those worsening after first dose.
Time Frame: Baseline up to 7-10 days after last dose of study drug (follow-up)
Population: All participants who received at least 1 dose of study drug were included in the AE summarization/analysis.
Measure: Number; unit: participants
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 82 | 80
participants
  Participants with TEAEs | 41 | 53 | 51
  Participants with SAEs | 2 | 0 | 6
  Participants discontinued permanently due to AEs | 2 | 9 | 8

9. Secondary Outcome: Number of Participants With Change From Baseline and Absolute Values in Vital Signs Meeting Categorical Summarization Criteria
Description: Categorical summarization criteria in vital signs included: sitting, supine, and standing systolic blood pressure (SBP) of less than (<)90 millimeters of mercury (mm Hg) or change in sitting, supine and standing SBP of more than or equal to (>=)30 mm Hg; supine, sitting, and standing diastolic blood pressure (DBP) of <50 mm Hg or change in sitting, supine, and standing DBP of >=20 mm Hg; supine and sitting pulse rate of <40 or more than (>)120 beats per minute (bpm); and standing pulse rate of <40 or >140 bpm.
Time Frame: Screening up to 7-10 days after last dose of study drug (follow-up)
Population: All participants who received at least 1 dose of study drug were included in the safety analyses. n=number of evaluable participants for each specified vital sign parameter.
Measure: Number; unit: participants
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 82 | 80
participants
  Supine SBP <90 mmHg (n=78,82,80) | 0 | 0 | 0
  Sitting SBP <90 mmHg (n=74,79,79) | 0 | 1 | 1
  Standing SBP <90 mmHg (n=78,82,80) | 0 | 2 | 1
  Supine DBP <50 mmHg (n=78,82,80) | 0 | 1 | 0
  Sitting DBP <50 mmHg (n=74,79,79) | 0 | 0 | 0
  Standing DBP <50 mmHg (n=78,82,80) | 0 | 0 | 0
  Supine pulse rate <40 or >120 bpm (n=78,82,80) | 0 | 0 | 0
  Sitting pulse rate <40 or >120 bpm (n=74,79,79) | 0 | 0 | 0
  Standing pulse rate <40 bpm (n=78,82,80) | 0 | 1 | 0
  Standing pulse rate >140 bpm (n=78,82,80) | 0 | 0 | 0
  Increase in supine SBP >=30 mmHg (n=75,81,79) | 3 | 1 | 3
  Increase in sitting SBP >=30 mmHg (n=73,79,79) | 0 | 2 | 2
  Increase in standing SBP >=30 mmHg (n=75,81,79) | 3 | 2 | 2
  Increase in supine DBP >=20 mmHg (n=75,81,79) | 3 | 1 | 4
  Increase in sitting DBP >=20 mmHg (n=73,79,79) | 2 | 2 | 5
  Increase in standing DBP >=20 mmHg (n=75,81,79) | 6 | 2 | 1
  Decrease in supine SBP >=30 mmHg (n=75,81,79) | 1 | 4 | 1
  Decrease in sitting SBP >=30 mmHg (n=73,79,79) | 2 | 2 | 2
  Decrease in standing SBP >=30 mmHg (n=75,81,79) | 1 | 2 | 1
  Decrease in supine DBP >=20 mmHg (n=75,81,79) | 3 | 0 | 3
  Decrease in sitting DBP >=20 mmHg (n=73,79,79) | 3 | 8 | 2
  Decrease in standing DBP >=20 mmHg (n=75,81,79) | 4 | 0 | 3

10. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Values Meeting Categorical Summarization Criteria
Description: Criteria for ECG (12-lead) values meeting categorical summarization criteria were: the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization (PR interval >=300 milliseconds (msec) and increase from baseline >=25/50%; time from the beginning of the electrocardiogram Q wave to the end of the S wave corresponding to ventricular depolarization (QRS) interval >=140 msec and increase of >=50%; the beginning of the Q wave to the end of the T wave corresponding to electrical systole (QT) interval corrected using the Fridericia formula (QTcF) of 450 to <480 msec, 480 to <500 msec and >=500 msec, or an increase of 30 to <60 msec or >=60 msec.
Time Frame: Screening/Baseline up to Week 12 (or Early Termination)
Population: All participants who received at least 1 dose of study drug were included in the safety analyses. n=number of evaluable participants for each specified ECG parameter.
Measure: Number; unit: participants
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 82 | 80
participants
  PR interval >=300 msec (n=78,82,80) | 0 | 0 | 0
  QRS >=140 msec (n=78,82,80) | 1 | 0 | 0
  QTcF 450 to <480 msec (n=78,82,80) | 5 | 6 | 2
  QTcF >=500 msec (n=78,82,80) | 0 | 0 | 0
  PR interval increase >=25/50% (n=72,81,77) | 0 | 0 | 0
  QRS increase >=50% (n=72,81,77) | 1 | 0 | 0
  QTcF increase 30 to <60 msec (n=72,81,77) | 3 | 1 | 3
  QTcF increase >=60 msec (n=72,81,77) | 0 | 0 | 1
  QTcF 480 to <500 msec (n=78,82,80) | 0 | 0 | 1

11. Secondary Outcome: Number of Participants With Weight Change >=7%
Description: The effects of PF-02545920 on body weight were evaluated. The number of participants with changes from baseline in body weight of >=7% were tabulated and summarized.
Time Frame: Screening up to Day 84
Population: All participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 82 | 80
participants
  Increase from baseline >=7% | 2 | 1 | 3
  Decrease from baseline >=7% | 1 | 7 | 3

12. Secondary Outcome: Number of Participants With New/Intensified Physical Examination Findings From Baseline by Body Site
Description: A complete physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems.
Time Frame: Baseline and Week 12 or Early Termination
Population: All participants who received at least 1 dose of study drug and who were evaluable for physical examinations.
Measure: Number; unit: participants
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 72 | 77 | 74
participants
  Ears | 0 | 0 | 0
  Eyes | 1 | 0 | 0
  Gastrointestinal | 0 | 0 | 1
  General Appearance | 1 | 0 | 1
  Head | 1 | 0 | 1
  Heart | 0 | 1 | 0
  Lungs | 0 | 0 | 0
  Lymph nodes | 0 | 0 | 0
  Mouth | 0 | 1 | 1
  Musculoskeletal | 2 | 1 | 0
  Neurological | 0 | 0 | 1
  Nose | 0 | 0 | 0
  Skin | 1 | 0 | 0

13. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Number of participants with laboratory test abnormalities without regard to baseline abnormality. Laboratory test parameters included hematology, liver function, renal function, lipids, electrolytes, hormones (prolactin), clinical chemistry, and urinalysis (dipstick and microscopy).
Time Frame: Screening up to Week 12/Early Termination and 7-10 days after last dose of study drug (hematology only)
Population: All participants who had received at least 1 dose of study drug and who were evaluable for laboratory abnormalities.
Measure: Number; unit: participants
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 75 | 81 | 78
participants | 46 | 54 | 49

14. Secondary Outcome: Number of Participants With Extrapyramidal Motor System (EPS) AEs
Description: EPS AEs consisted of oromandibular dystonia, extrapyramidal disorder, akathisia, dyskinesia, and tremor.
Time Frame: Baseline up to 7-10 days after last dose of study drug (follow-up)
Population: All participants who received at least 1 dose of study drug were included in the AE summarization/analysis.
Measure: Number; unit: participants
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 82 | 80
participants
  Oromandibular dystonia | 0 | 2 | 0
  Extrapyramidal disorder | 0 | 1 | 0
  Akathisia | 0 | 2 | 0
  Dyskinesia | 0 | 2 | 0
  Tremor | 0 | 3 | 0

15. Secondary Outcome: Change From Baseline in Cholesterol, Triglycerides (TG), Low-Density Lipoprotein (LDL), and High-Density Lipoprotein (HDL) at Weeks 6 and 12
Description: Choleseterol, TG, glycosylated hemoglobin (HbA1c), LDL, HDL, insulin, and prolactin were a part of the laboratory tests done (metabolic tests).
Time Frame: Baseline; Weeks 6 and 12
Population: All participants who had received at least 1 dose of study drug and who had available data for metabolic parameters. n=number of evaluable participants at the specified time points.
Measure: Mean (Standard Deviation); unit: milligram (mg)/deciliter (dL)
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 81 | 78
milligram (mg)/deciliter (dL)
  Cholesterol, baseline (n=78,81,78) | 197.4 (41.84) | 196.9 (39.08) | 188.6 (42.42)
  Cholesterol, change at Week 6 (n=53,45,58) | -2.5 (25.03) | -6.2 (24.89) | -1.1 (22.82)
  Cholesterol, change at Week 12 (n=71,67,65) | -5.3 (31.56) | -8.9 (25.49) | 0.3 (24.38)
  TG, baseline (n=78,81,78) | 126.7 (82.31) | 125.3 (62.13) | 143.0 (121.41)
  TG, change at Week 6 (n=53,45,58) | 7.7 (69.01) | -15.0 (59.10) | 3.1 (68.39)
  TG, change at Week 12 (n=71,67,65) | -3.7 (57.77) | -10.2 (60.46) | 7.8 (67.02)
  LDL, baseline (n=77,81,76) | 113.6 (34.80) | 115.1 (35.22) | 108.3 (31.88)
  LDL, change at Week 6 (n=52,45,56) | -1.5 (19.19) | -1.1 (21.97) | -1.5 (19.57)
  LDL, change at Week 12 (n=70,67,61) | -2.8 (24.29) | -7.3 (20.87) | 0.5 (20.88)
  HDL, baseline (n=78,81,78) | 57.8 (19.06) | 56.7 (15.17) | 51.5 (13.28)
  HDL, change at Week 6 (n=53,45,58) | -2.7 (8.71) | -2.1 (8.41) | -0.2 (5.83)
  HDL, change at Week 12 (n=71,67,65) | -1.5 (10.22) | 0.5 (7.46) | 0.8 (7.26)

16. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Weeks 6 and 12
Description: Choleseterol, TG, HbA1c, LDL, HDL, insulin, and prolactin were a part of the laboratory tests done (metabolic tests).
Time Frame: Baseline; Weeks 6 and 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 81 | 78
percent
  Baseline (n=78,81,77) | 5.70 (0.638) | 5.74 (0.619) | 5.70 (0.651)
  Change at Week 6 (n=53,45,58) | -0.04 (0.321) | 0.00 (0.234) | 0.01 (0.290)
  Change at Week 12 (n=70,67,65) | -0.05 (0.278) | -0.07 (0.305) | -0.07 (0.314)

17. Secondary Outcome: Change From Baseline in Insulin at Weeks 6 and 12
Description: Choleseterol, TG, HbA1c, LDL, HDL, insulin, and prolactin were a part of the laboratory tests done (metabolic tests).
Time Frame: Baseline; Weeks 6 and 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: micro international unit/milliliter
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 81 | 78
micro international unit/milliliter
  Baseline (n=74,80,78) | 9.19 (7.907) | 9.78 (8.902) | 9.53 (7.575)
  Change at Week 6 (n=48,48,62) | 4.94 (16.755) | 3.04 (16.933) | 3.02 (14.157)
  Change at Week 12 (n=67,67,69) | 7.40 (26.838) | 1.29 (9.230) | 1.30 (9.399)

18. Secondary Outcome: Change From Baseline in Prolactin at Weeks 6 and 12
Description: Choleseterol, TG, HbA1c, LDL, HDL, insulin, and prolactin were a part of the laboratory tests done (metabolic tests).
Time Frame: Baseline; Weeks 6 and 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: nanogram (ng)/milliliter
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 81 | 78
nanogram (ng)/milliliter
  Baseline (n=78,81,77) | 13.71 (18.954) | 13.29 (17.709) | 12.51 (13.597)
  Change at Week 6 (n=52,45,57) | 0.27 (6.410) | 2.65 (12.080) | 0.99 (9.074)
  Change at Week 12 (n=70,68,64) | 0.04 (8.834) | 2.65 (15.786) | 0.01 (8.925)

19. Secondary Outcome: Change From Baseline to Week 12 on the Extrapyramidal Symptom Rating Scale-Abbreviated (ESRS-A)
Description: The ESRS-A is a 28-item instrument designed to facilitate standardized observations of parkinsonism, dystonia, dyskinesia, and akathisia. Ratings were determined through a combination of clinical interview and a motor examination. Scores were divided into individual domain scores and clinical global impression scores (CGI-S). Scores started from 0 (normal) to 6 (0 to 8 for CGI-S), with higher scores indicating greater severity.
Time Frame: Baseline, Week 12
Population: All participants who received at least 1 dose of study drug. n=number of evaluable participants for each parameter at the specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 82 | 80
units on a scale
  Parkinsonism, baseline (n=78,82,80) | 0.5 (1.70) | 0.8 (1.82) | 0.2 (0.69)
  Parkinsonism, change at Week 12 (W12) (n=43,38,53) | -0.3 (1.77) | 0.1 (2.01) | -0.0 (0.44)
  Dystonia, baseline (n=78,82,80) | 0.1 (0.27) | 0.0 (0.00) | 0.0 (0.11)
  Dystonia, change at W12 (n=43,38,53) | -0.0 (0.21) | 0.1 (0.23) | 0.0 (0.00)
  Dyskinesia, baseline (n=78,82,80) | 0.1 (0.50) | 0.1 (0.46) | 0.2 (0.62)
  Dyskinesia, change at W12 (n=43,38,53) | -0.0 (0.21) | 0.0 (0.00) | 0.2 (0.66)
  Akathisia, baseline (n=78,82,80) | 0.3 (0.87) | 0.3 (0.68) | 0.2 (0.83)
  Akathisia, change at W12 (n=43,38,53) | -0.1 (0.54) | 0.0 (0.97) | -0.1 (1.02)
  CGI-S Parkinsonism, baseline (n=78,82,80) | 0.2 (0.45) | 0.3 (0.68) | 0.1 (0.33)
  CGI-S Parkinsonism, change at W12 (n=43,38,53) | -0.1 (0.34) | 0.1 (0.73) | 0.0 (0.20)
  CGI-S Dystonia, baseline (n=78,82,80) | 0.1 (0.25) | 0.0 (0.00) | 0.0 (0.11)
  CGI-S Dystonia, change at W12 (n=43,38,53) | -0.1 (0.26) | 0.0 (0.16) | 0.0 (0.20)
  CGI-S Dyskinesia, baseline (n=78,82,80) | 0.1 (0.27) | 0.1 (0.29) | 0.1 (0.39)
  CGI-S Dyskinesia, change at W12 (n=43,38,53) | -0.0 (0.15) | 0.0 (0.00) | 0.1 (0.41)
  CGI-S Akathisia, baseline (n=78,82,80) | 0.2 (0.46) | 0.1 (0.35) | 0.1 (0.43)
  CGI-S Akathisia, change at W12 (n=43,38,53) | -0.1 (0.37) | -0.0 (0.54) | -0.1 (0.53)

20. Secondary Outcome: Absolute Values of Movement Disorder Burden Score - Dystonia (MDBS-D) Over Active Treatment Period
Description: The MDBS-D quantified the dystonia burden during the active treatment period. For an individual participant, MDBS-D took into account all treatment-emergent dystonia events and was defined as a combination of the severity of the AE due to dystonia, AE duration, prescribed concomitant medication, and the total number of days the study treatment was received. Scores for the MDBS-D ranged from 0 (no dystonia events) to 4.5, with higher scores indicating greater dystonia burden.
Time Frame: Active treatment period (Weeks 1 to 12/Early Termination)
Population: All participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 82 | 80
units on a scale | 0.00 (0.000) | 0.02 (0.175) | 0.00 (0.000)

21. Secondary Outcome: Overall Number of Participants With Positive Responses to Categories on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS assessed whether participant experienced the following: completed suicide (Category 1), suicide attempt (Category 2; response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (Category 3; "Yes" on "preparatory acts or behavior"), suicidal ideation (Category 4; "Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent), any suicidal behavior or ideation, self-injurious behavior (Category 7; "Yes" on "Has subject engaged in non-suicidal self-injurious behavior").
Time Frame: Baseline up to 7-10 days after last dose of study drug
Population: All participants who had received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 78 | 82 | 80
participants
  Category 1 | 0 | 0 | 0
  Category 2 | 0 | 0 | 0
  Category 3 | 0 | 0 | 0
  Category 4 | 1 | 3 | 1
  Category 7 | 0 | 0 | 0

22. Secondary Outcome: Concentration of PF-02545920 and Its Metabolite, PF-01001252
Description: Pharmacokinetic (PK) samples were collected at varying times relative to drug dosing whenever participants could be scheduled for study visits (sparse PK sampling). Thus, because of the variable time between the last dose and the collection of the PK samples, typical summary PK analyses were not planned or described in the study protocol and are not available. The study protocol analysis section specified that the sparse sampled PK data might be pooled with PK data from previous PF-02545920 clinical studies, however the study results did not support conducting those analyses.
Time Frame: Days 14, 28, 42, 56, 70, 84/Early Termination
Population: Summary PK analyses were not planned or performed due to sparse PK sampling.
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: All treated participants were analyzed for AEs. The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-02545920 5 mg BID | PF-02545920 15 mg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 2/78 | 0/82 | 6/80
Other Adverse Events (participants affected / at risk) | 20/78 | 22/82 | 25/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-02545920 5 mg BID (N=78) | PF-02545920 15 mg BID (N=82) | Placebo (N=80)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Paranoia (Psychiatric disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-02545920 5 mg BID (N=78) | PF-02545920 15 mg BID (N=82) | Placebo (N=80)
Dry mouth (Gastrointestinal disorders) | 4 | 4 | 3
Nausea (Gastrointestinal disorders) | 2 | 4 | 5
Vomiting (Gastrointestinal disorders) | 4 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 6
Headache (Nervous system disorders) | 5 | 1 | 6
Sedation (Nervous system disorders) | 4 | 6 | 7
Somnolence (Nervous system disorders) | 5 | 8 | 2

LIMITATIONS AND CAVEATS:
The study was terminated prematurely as a pre-planned interim analysis indicated the study was unlikely to meet the pre-specified efficacy criteria. The decision was not based on any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.